CLINICAL TRIAL: NCT03017521
Title: A Phase II Study of TAS-117 in Advanced Solid Tumors With PI3K/AKT Gene Aberration (Part of K-BASKET Trial; Korea-Biomarker-driven Multi-arm Drug-screening, Knowledge and Evidence-generating Targeted Trial)
Brief Title: K-BASKET, TAS-117, PI3K/AKT Gene Aberration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Minkyu Jung, Assistant Professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2016-0743
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Solid Tumor, Adult
Keywords: Refractory solid tumors; AKT inhibitor
MeSH Terms: interventions — 3-amino-1-methyl-3-(4-(3-phenyl-5H- imidazo(1,2-c)pyrido(3,4-e)(1,3)oxazin-2-yl)phenyl)cyclobutanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAS-117 (Experimental): TAS-117, 16mg, orally, daily
  Interventions: Drug: TAS-117

INTERVENTIONS:
Drug: TAS-117 — TAS-117 16mg, daily

SUMMARY:
The phosphatidylinositol 3-kinase (PI3K)-v-akt murine thymoma viral oncogene homolog (AKT)-mammalian target of rapamycin (mTOR) signaling pathway is one of the most frequently aberrantly regulated pathways in human tumors. TAS-117 is a highly potent and selective oral allosteric AKT inhibitor. It has high affinity for AKT1, 2, and 3 and shows potent anti-proliferative activity against multiple tumor cell lines in vivo. Therefore, we propose to conduct a phase II trial of TAS-117, potent and selective AKT inhibitor, in patients with advanced solid tumor with PI3K/AKT genetic aberrancy by NGS focusing panel in part of K-BASKET trial.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed recurrent or advanced solid cancers with PI3K/ATK aberration
2. Progressive disease who failed to previous standard treatment.
3. At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors version 1.1 criteria
4. Eastern Cooperative Oncology Group performance status 0 or 1
5. Able to take medications orally
6. Adequate organ function
7. A life expectancy of at least 60 days

Exclusion Criteria:

1. Previous treatment with anti-PI3K or AKT directed therapies
2. Known hypersensitivity to any drugs similar to TAS-117 in structure or class.
3. History or current evidence of type 1 or type 2 diabetes mellitus that requires insulin and/or oral antidiabetic therapy.
4. Current evidence of retinopathy that requires ophthalmological therapy.
5. History or current evidence of cardiac arrhythmia and/or conduction abnormality.
6. Treatment with any of the following within the specified time frame prior to study drug administration:

   * Major surgery within prior 4 weeks
   * Radiation therapy for extended field within 4 weeks prior to study drug administration or limited field radiation therapy within 2 weeks prior to study drug administration.
   * Any anticancer treatment within 3 weeks prior to study drug administration (mitomycin within prior 5 weeks).
7. A serious illness or medical condition(s)
8. Unresolved toxicity of Grade >1 attributed to any prior therapies (excluding alopecia, skin pigmentation and anemia).
9. Patients with the risk of hypokalemia
10. Receiving oral steroid medication.
11. Pregnant or lactating female

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
overall response rate | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee JB, Jung M, Beom SH, Kim GM, Kim HR, Choi HJ, Sohn JH, Ahn JB, Rha SY, Chung HC. Phase 2 study of TAS-117, an allosteric akt inhibitor in advanced solid tumors harboring phosphatidylinositol 3-kinase/v-akt murine thymoma viral oncogene homolog gene mutations. Invest New Drugs. 2021 Oct;39(5):1366-1374. doi: 10.1007/s10637-021-01085-7. Epub 2021 Mar 15. PMID 33723724